CLINICAL TRIAL: NCT04379817
Title: Somatostatin Receptors Imaging in Relapsing and Refractory Multiple Myeloma Patients
Acronym: SCARLET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IJBMNSSTR
Record Dates: First submitted 2020-04-14; First posted 2020-05-08 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2023-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gallium-68 labelled DOTA-conjugated SSTR targeting peptide PET/CT — Assess somatostatin receptor expression

SUMMARY:
This study wil assess somatostatin receptor (SSTR) expression via the uptake of Gallium-68 labelled DOTA-conjugated SSTR targeting peptide using PET/CT imaging in multiple myeloma lesions pre-identified on 18F-FDG PET/CT in order to evaluate the feasibility of molecular radionuclide therapy in refractory and relapsing mutiple myeloma using the Lutetium-177 radiolabelled targeting peptide.

ELIGIBILITY:
Inclusion Criteria:

* Age above or equal to 18 years
* Written informed consent in accordance with institutional guidelines and obtained prior to any study procedures
* Confirmed diagnosis of multiple myeloma according to the Salmon and Durie criteria
* Has received at least 3 lines of treatment, exposed and refractory (or non-eligible) to the 5 major drugs (lenalidomid, pomalidomid, bortezomib, carfilzomib, daratumumab)
* Life expectancy above 3 months
* Active (relapsing or refractory) and measurable disease (on 18F-FDG PET/CT (performed within 4 weeks prior SSTR PET/CT) and biologically)
* Adequate renal function with GFR above or equal to 30mL/min/1.73m²
* Bone marrow aspiration and biopsy sample available within 30 days prior study enrolment with positive SSTR2 IHC

Exclusion Criteria:

* Pregnant or lactating patients
* Other active neoplastic disease
* Treatment by another molecule that is object of investigation within 30 days prior SSTR PET/CT
* Eastern Cooperative Oncology Group Performance Status above or equal to 3
* Corticoids administration at a therapeutic level (total dose of 160 mg of dexamethasone or equivalent) two weeks prior enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Somatostatin receptor expression | through study completion, an average of 1,5 year
  Biodistribution of 68Ga-DOTA cojugated SSTR targeting peptide on PET/CT images

CONTACTS AND LOCATIONS:
Locations (1):
- Jules Bordet Institute, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delbart W, Karfis I, Vercruyssen M, De Wind R, Meuleman N, Wimana Z, Flamen P, Woff E. The SCARLET trial: a prospective phase II study of somatostatin receptor imaging for potential radiotheranostic application in patients with relapsing and refractory multiple myeloma. Eur J Nucl Med Mol Imaging. 2026 Feb;53(3):1521-1531. doi: 10.1007/s00259-025-07500-y. Epub 2025 Aug 28. PMID 40866646